CLINICAL TRIAL: NCT05690074
Title: Monitoring the Effect of Epidural Stimulation on Sensorimotor and Autonomic Functions in Chronic Patients With Spinal Cord Injury
Brief Title: Epidural Stimulation in Chronic Spinal Cord Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Vojtech Rybka, MD, Principal Investigator, University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK-1302/21
Record Dates: First submitted 2022-12-02; First posted 2023-01-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; spinal cord stimulation; volitional movement; functional magnetic resonance imaging; autonomic nervous system
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with chronic spinal cord injury (Experimental): 80 sessions each of epidural spinal cord stimulation for 1) autonomic functions 2) voluntary movement; and 3) standing
  Interventions: Device: Spectra Wave Writer™ Spinal Cord Stimulator System

INTERVENTIONS:
Device: Spectra Wave Writer™ Spinal Cord Stimulator System — Device: 5-6-5 Specify electrode Device: Restore Advance Pulse Generator

SUMMARY:
Investigators propose to demonstrate that epidural stimulation (ES) can be used to recover significant levels of autonomic control of cardiovascular, urinary and sexual function as well as the ability to voluntarily control leg movements below the injury level. This intervention would provide an immediate therapeutic alternative to individuals who now have no recourse for treatment. In addition investigators suggest to prove on functional magnetic resonance imaging if there are some significant changes before and after the stimulation.

ELIGIBILITY:
Inclusion Criteria:

* non-progressive SCI with complete motor paralysis below T1; American Spinal Injury Association Impairment Scale (AIS) A or B
* 18 - 60 years of age;
* longer than 2 years post injury;
* stable medical condition
* unable to voluntarily move all single joints of the legs;
* spinal cort lesion between C7 and Th10

Exclusion Criteria:

* ventilator dependent;
* painful musculoskeletal dysfunction, unhealed fracture, contracture, or pressure sore that might interfere with training;
* clinically significant depression or ongoing drug abuse;
* cardiovascular, respiratory, bladder, or renal disease unrelated to SCI;
* severe anemia (Hgb<8 g/dl) or hypovolemia; and HIV or AIDS related illness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Brain functional connectivity | 1 year after implantation
  Researchers want to describe if there are some changes on functional MRI of the spinal cord and brain before and after stimulation. With functional MRI in rest and task condition, the functional connectivity (FC) is examined.
Change from baseline of lower extremity independence time during after 1 year of stimulation | 1 year after stimulation (360 training sessions)
  Researchers will measure the amount of time individuals are able to stand without manual assistance (independently).

SECONDARY OUTCOMES:
Change in trunk stability restoration | 6 month and 1 year after implantation
  Trunk control stability test in individuals with spinal cord injury (SCI)
Neurogenic bladder symptoms will be measured using the Neurogenic Bladder Symptom Score (NBSS). | 3 month, 6 month, 9 month, 12 month
  Assessment of neurogenic bladder symptoms will be performed to assess the impact of long term eSCS on this measure. The score measures bladder symptoms across 3 different domains: incontinence (scored 0-29), storage and voiding (scored 0-22), and consequences (scored 0-23), with higher scores representing worse symptoms.
Sexual function as measured by the Sexual Function Questionnaire | 3 month, 6 month, 9 month, 12 month
  The Sexual Function Questionnaire (SFQ) is a self-report outcome measure of sexual function.
Change in sense of wellbeing as measured by the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire | 3 month, 6 month, 9 month, 12 month
  The WHOQOL-BREF assesses quality of life (QOL) within the context of an individual's culture, value systems, personal goals, standards and concerns. The higher score in the questionnaire means better quality of life for patient.
Symptoms of spasticity will be measured by Modified Ashworth spasticity test | 3 month, 6 month, 9 month, 12 month
  The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone.
Neurogenic bowel symptoms will be measured using the Neurogenic Bowel Dysfunction (NBD) score. | 3 month, 6 month, 9 month, 12 month
  Assessment of neurogenic bowel symptoms will be performed to assess the impact of long term eSCS on this measure. Scores can range from 0-47, with a higher score representing more severe dysfunction.
Reduction of neuropathic pain | 3 month, 6 month, 9 month, 12 month
  We will measure neuropathic pain by the Neuropathic Pain Questionnaire (NPQ)
Change in BP during the head up tilt test (HUTT) | 6 month -1 year
  During HUTT, participants will be passively moved to approximately 60° upright stand position by the investigators using the tilt table. Using epidural spinal cord stimulation (eSCS) to activate spinal sympathetic circuitry and mitigate low resting BP and orthostatic hypotension (OH) and continuous beat-by beat BP monitoring via finger photoplethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Kriz, MD, PhD, Study Chair — UH Motol - spinal cord unit
Locations (1):
- UH Motol, Prague, Czechia

REFERENCES:
- [Background] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Background] Harkema S, Gerasimenko Y, Hodes J, Burdick J, Angeli C, Chen Y, Ferreira C, Willhite A, Rejc E, Grossman RG, Edgerton VR. Effect of epidural stimulation of the lumbosacral spinal cord on voluntary movement, standing, and assisted stepping after motor complete paraplegia: a case study. Lancet. 2011 Jun 4;377(9781):1938-47. doi: 10.1016/S0140-6736(11)60547-3. Epub 2011 May 19. PMID 21601270
- [Background] Gerasimenko YP, Lu DC, Modaber M, Zdunowski S, Gad P, Sayenko DG, Morikawa E, Haakana P, Ferguson AR, Roy RR, Edgerton VR. Noninvasive Reactivation of Motor Descending Control after Paralysis. J Neurotrauma. 2015 Dec 15;32(24):1968-80. doi: 10.1089/neu.2015.4008. Epub 2015 Aug 20. PMID 26077679
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Zhang H, Liu Y, Zhou K, Wei W, Liu Y. Restoring Sensorimotor Function Through Neuromodulation After Spinal Cord Injury: Progress and Remaining Challenges. Front Neurosci. 2021 Oct 14;15:749465. doi: 10.3389/fnins.2021.749465. eCollection 2021. PMID 34720867
- [Background] Choi EH, Gattas S, Brown NJ, Hong JD, Limbo JN, Chan AY, Oh MY. Epidural electrical stimulation for spinal cord injury. Neural Regen Res. 2021 Dec;16(12):2367-2375. doi: 10.4103/1673-5374.313017. PMID 33907008
- [Background] Pena Pino I, Hoover C, Venkatesh S, Ahmadi A, Sturtevant D, Patrick N, Freeman D, Parr A, Samadani U, Balser D, Krassioukov A, Phillips A, Netoff TI, Darrow D. Long-Term Spinal Cord Stimulation After Chronic Complete Spinal Cord Injury Enables Volitional Movement in the Absence of Stimulation. Front Syst Neurosci. 2020 Jun 30;14:35. doi: 10.3389/fnsys.2020.00035. eCollection 2020. PMID 32714156